CLINICAL TRIAL: NCT05280691
Title: A Multi-center, Cluster Randomized Superiority Trial of a Guideline-based Family Support Intervention in Intensive Care Units
Brief Title: Family Support Intervention in Intensive Care Units
Acronym: FICUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rahel Naef (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor-Investigator, Rahel Naef, Assistant Professor of Implementation Science in Nursing, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0001
Record Dates: First submitted 2022-02-20; First posted 2022-03-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Postintensive Care Syndrome; Family Members; Quality of Life; Depression, Anxiety; Posttraumatic Stress Disorder; Family Dynamics
Keywords: Family illness management; Family support intervention
MeSH Terms: conditions — postintensive care syndrome; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The trial is designed as a multi-center, parallel-cluster randomized, superiority trial with 16 clusters of ICUs in the German-speaking part of Switzerland.
  The study aims to determine the effect of a nurse-led, interprofessional family support intervention on quality of family care, family management, and individual mental health compared to usual care provided to family members. The study also aims to identify implementation barriers/enablers in the real-world context in which the study intervention is implemented to discern determinants and strategies of implementation success.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family Support Intervention (Other): Families in the intervention group receive the Family Support Intervention in addition to usual care
  Interventions: Other: Family Support Intervention (FSI)
- Usual Care (No Intervention): Families in the control group will receive usual care.

INTERVENTIONS:
Other: Family Support Intervention (FSI) — In addition to usual care, families in the intervention group will receive (1) specialist nurse support along the patient pathway at defined time-points, from admission to discharge including follow-up care, and (2) nurse-coordinated liaison and structured, interprofessional communication by the ICU team. The intervention is grounded in a family systems approach and guideline-based strategies for family engagement in the ICU and has been pilot-tested in one ICU.
  Arms: Family Support Intervention

SUMMARY:
Background: Family members of critically ill patients face considerable uncertainty and distress during their close other's intensive care unit (ICU) stay, with about 20-60% of family members experiencing post-traumatic distress post-ICU. Guidelines recommend structured family inclusion, communication, and support, but the existing evidence base around protocolized family support interventions is modest and requires substantiation.

Methods: To test the clinical effectiveness and explore the implementation of a multicomponent, nurse-led family support intervention in ICUs, the investigators will undertake a parallel, cluster-randomized, controlled, multicenter superiority hybrid-type 1 trial. The trial will include eight clusters (ICUs) per study arm, with a projected total sample size of 896 family members of adult, critically ill patients treated in the German-speaking part of Switzerland. The trial targets family members of critically ill patients with an expected ICU stay of 48 hours or longer. Families in the control arm will receive usual care. Families in the intervention arm, in addition to usual care, will receive a family support intervention consisting of specialist nurse support along the patient pathway at defined time-points, including follow-up care, and nurse-coordinated liaison and structured, interprofessional communication by the ICU team. The primary study endpoint is quality of family care, operationalized as family members' satisfaction with ICU care at discharge. Secondary endpoints include quality of communication and nurse support, family management of critical illness (functioning, resilience), and family members' mental health (well-being, psychological distress) measured at admission, discharge, and after three, six, and twelve months. Data of all participants, regardless of protocol adherence, will be analyzed using linear mixed-effects models, with the individual participant as the unit of inference.

Discussion: The FICUS trial will establish the effectiveness of the family support intervention and generate knowledge of its implementability. Both types of evidence are necessary to determine whether the intervention works as intended in clinical practice and whether an effective intervention could be scaled-up to other ICUs. The study findings will make a significant contribution to the current body of knowledge on effective ICU care that promotes family participation and well-being.

DETAILED DESCRIPTION:
Background: Family members are important to the well-being and recovery of critically ill persons, yet are themselves profoundly affected by the critical illness. During a close other's treatment in an intensive care unit (ICU), families experience high levels of stress and uncertainty, particularly in the event of surrogate decision-making and loss. Poor communication, insufficient shared decision-making, and inadequate emotional and practical support by intensive care staff have been found to add to families' burden. Poor-quality care has been associated with adverse mental health outcomes, which is reported by 20-60% of family members. A lack of engagement and support, coupled with acute stress, not only increases family suffering, but affects family members' functioning in everyday life, and limits their ability to engage in caregiving activities needed by the survivor of critical illness or cope with their loss.

Rationale: To increase the quality of family care and prevent adverse mental health outcomes, ICU guidelines recommend family engagement, communication, and support as well as the use of specific roles, but the evidence base for these recommendations is weak to date. Only a few studies have investigated family support interventions that consist of structured communication and / or specific family nursing roles. Promising effects have been found on family members' communication and support experience. However, findings on psychological distress remain inconclusive whereas insights on family management ability are virtually absent. Moreover, best practice around family engagement in ICU is often not implemented consistently in routine care. Hence, real-world evidence generated by randomized controlled designs is necessary to establish the effect of such multi-component interventions on quality of family care and their potential in supporting family management of critical illness and in reducing adverse mental health outcomes.

Aims: The study aims to determine the effect of a guideline-based, nurse-led, interprofessional family support intervention on quality of family care, family management, and individual mental health compared to usual care provided to family members. The study also aims to identify implementation barriers/enablers in the real-world context in which the study intervention is implemented to discern determinants and strategies of implementation success.

Methodology: The trial is designed as a multi-center, parallel cluster randomized superiority hybrid-type 1 trial with 8 clusters per study arm and a projected sample size of 896 family members of adult, critically ill patients treated in acute care hospitals in the German-speaking part of Switzerland. It will target family members with great needs, such as those of patients with more complex and longer-lasting critical illness, those of patients admitted with a life-threatening condition, and those who are required to make surrogate decisions. Family members of patients requiring short-lasting peri-operative or peri-interventional ICU treatment will be excluded. In addition to usual care, families in the intervention group will receive (1) specialist nurse support along the patient pathway at defined time-points, from admission to discharge with subsequent follow-up care, and (2) nurse-coordinated liaison and structured, interprofessional communication by the ICU team. Family members in the control group will receive usual care. The primary study endpoint is quality of family care, operationalized as family members' satisfaction with ICU care at discharge. Secondary endpoints include quality of communication and nurse support, family management of critical illness (functioning, resilience), and index family members' mental health (well-being, psychological distress) obtained upon admission, discharge, and after 3, 6, and 12 months. Data of all participants, regardless of protocol adherence, will be analyzed using linear mixed-effects models, with the individual participant as the unit of inference. A mixed-method study will be used to examine implementation barriers / facilitators and successful strategies at intervention units.

Expected outcomes and impact: The FICUS trial will establish the effectiveness of the family support intervention and generate knowledge on effective implementation processes. Both types of evidence are necessary to determine whether the intervention works as intended, but also to explore how it works in clinical practice, so that an effective intervention could be scaled-up to other ICUs. The study findings will make a significant contribution to the current body of knowledge on effective ICU care that promotes family participation and well-being. They will also promote evidence-based family care in ICU.

ELIGIBILITY:
Potential participants are family members of critically ill persons admitted to a study ICU. A family member is defined as a close other from the patient's perspective, as noted in the clinical record or in advanced directives, or as indicated by the legally defined surrogate decision-maker.

Inclusion criteria regarding patients (one or several):

* Expected length of stay in ICU ≥48 hours, as predicted by the intaking ICU clinician (physician or nurse) at admission.
* Life-threatening condition with a high risk of death or long-lasting functional impairment.
* High risk of prolonged mechanical ventilation (>24 hours).

Inclusion criteria regarding family members (all must apply):

* Primary support person of the patient.
* Able to complete family-reported outcome measures (questionnaires) in German language.
* Age ≥18 years.
* Signed informed consent form.

Exclusion criteria regarding patients (one leads to exclusion):

* Preexisting declined general consent.
* ICU stay <24 hours.

Exclusion criteria regarding family members (one leads to exclusion):

* Prior inclusion in FICUS trial on another study ICU.
* Cognitive inability to understand the study or complete the questionnaire as appraised by clinicians and / or study recruitment staff.
* Inability to complete baseline data collection within the required timeframe after admission / study enrollment (Calvert et al., 2018).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Care (Quality of Family Care) | Assessed no earlier than 24 hours prior to and no later than 14 days following the discharge of the patient from ICU.
  Quality of family care in ICU is operationalized as family satisfaction with ICU care, and measured with the Family Satisfaction in ICU questionnaire (FS-ICU-24R, German version). The FS-ICU-24R is a well-established instrument that assesses satisfaction with care (16 items) and satisfaction with involvement in decision-making (ten items). Its scores range from 0-100 with 100 indicating maximal satisfaction.

SECONDARY OUTCOMES:
Quality of Communication (Quality of Family Care) | Assessed no earlier than 24 hours prior to and no later than 14 days following the discharge of the patient from ICU.
  The Questionnaire on the Quality of Physician-Patient Interaction (QQPPI, original German version) is used to assess quality of communication between the ICU staff and family members during consultation. The 14 items assess aspects such as relationship-building, information exchange, and shared decision-making. The mean score ranges from 1-5 with a higher score indicating higher quality.
Nurse Support (Quality of Family Care) | Assessed no earlier than 24 hours prior to and no later than 14 days following the discharge of the patient from ICU.
  The Iceland Family Perceived Support Questionnaire (ICE-FPSQ, German version) is used to measure families' perception of support provided by nurses. The original English version has two subscales - emotional support (nine items) and cognitive support (five items). The ICE-FPSQ has been translated into German and is currently being validated prior to its use in the trial. A sum score is calculated for the total scale (range 14-70) and each subscale - emotional support (range 9-45) and cognitive support (range 5-25) - with higher scores indicating perception of better family support by nurses.
Family Functioning (Family Management) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  The Family Assessment Device - General Functioning Scale (FAD-GF-12, German version) - is used to assess overall functioning of the family system by six positive and six negative items. The mean score ranges from 1-4 with a lower score reflecting better functioning.
Family Resilience (Family Management) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  The Brief Resilience Scale (BRS, German version) measures the essence of resilience as the ability to bounce back from stress and is made up of three positive and three negative items. The items will be reformulated from "I" to "we" statements to assess the families' ability to bounce back from stress. The mean score ranges from 1-5 with a higher score indicating greater resilience.
Satisfaction with Life (Subjective Well-Being) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  The Satisfaction with Life Scale (SWLS-5, German version) measures the global dimension of subjective well-being. The sum score ranges from 5-35 with a higher score indicating a higher degree of satisfaction. It can be treated as an ordinal variable with seven levels using established thresholds.
Well-Being (Subjective Well-Being) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  The World Health Organization-5 Well-being Index (WHO-5, German version) measures subjective psychological well-being and is made up of five items tapping three major dimensions of positive affect as well as energy within the past two weeks. Its score ranges from 0-100, with a higher score indicating greater well-being, and has a threshold of 50 indicating depression.
Quality of Life (Subjective Well-Being) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  An adapted version of the general Quality of Life a Visual Analog Scale (QoL-VAS) as used in the EuroQol EQ-5D questionnaire will be employed to measure general rather than health-related quality of life. The score ranges from 0-100 with a higher score representing higher quality of life.
Psychological Distress (Mental Health) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  The Distress Thermometer (DT, German version) is a validated single-item screening instrument for distress in the past week originally (and still primarily) used among cancer patients with an established threshold for potential distress It ranges from 0-100 with a higher score indicating a higher level of distress.
Posttraumatic Stress (Mental Health) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  The Impact of Events Scale-R (IES-R) measures the presence and severity of symptoms associated with a traumatic event during the past week, and has three subscales - intrusion, avoidance, and hyperarousal. The six-item brief version (IES-6) used in this study includes two items from each of the three subscales, and its simple sum score (range 0-24 with a higher score indicating higher impact) has been shown to be highly correlated to the IES-R in various populations.
Depression, Anxiety (Mental Health) | Assessed within 96 hours after the admission of the patient to ICU, at the discharge from ICU (between 24 hours prior and 14 days after), 3 months (76-104 days), 6 months (166-194 days), and 12 months (351-379 days) after the discharge from ICU.
  The Hospital Anxiety and Depression Scale (HADS, German version) is made up of 14 items with different response categories scored in two subscales - anxiety (HADS-A, seven items) and depression (HADS-D, seven items) - and has thresholds for mild depression or anxiety and caseness for depression or anxiety, respectively. The scores range from 0-21 with a higher score indicating worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rahel Naef, PhD, RN, Principal Investigator — University of Zurich; Miodrag Filipovic, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Marie-Madlen Jeitziner, PhD, RN, Principal Investigator — University Hospital Bern, Inselspital
Locations (12):
- Switzerland (12):
  - Cantonal Hospital Winterthur, Winterthur, Canton of Zurich
  - Cantonal Hospital Baden, Baden
  - Lindenhof-Hospital, Bern
  - University Hospital Bern - Inselspital, Bern
  - Cantonal Hospital Graubünden, Chur
  - Spital Thurgau AG, Cantonal Hospital Frauenfeld, Frauenfeld
  - Lucerne Cantonal Hospital, Lucerne
  - Solothurn Hospitals AG, Cantonal Hospital Olten, Olten
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - Hospital Thun, Thun
  - University Hospital Zurich, Zurich
  - Hirslanden Clinic Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oesch S, Verweij L, Riguzzi M, Finch T, Naef R. Exploring Implementation Processes of a Multicomponent Family Support Intervention in Intensive Care Units (FICUS) Study: A Mixed-Methods Process Evaluation. J Adv Nurs. 2025 Nov;81(11):7245-7265. doi: 10.1111/jan.16544. Epub 2024 Oct 18. PMID 39422155
- [Background] Verweij L, Oesch S, Naef R. Tailored implementation of the FICUS multicomponent family support intervention in adult intensive care units: findings from a mixed methods contextual analysis. BMC Health Serv Res. 2023 Dec 1;23(1):1339. doi: 10.1186/s12913-023-10285-1. PMID 38041092
- [Background] Walker SP, Gaskin P, Powell CA, Bennett FI, Forrester TE, Grantham-McGregor S. The effects of birth weight and postnatal linear growth retardation on blood pressure at age 11-12 years. J Epidemiol Community Health. 2001 Jun;55(6):394-8. doi: 10.1136/jech.55.6.394. PMID 11350995
- [Background] Naef R, Filipovic M, Jeitziner MM, von Felten S, Safford J, Riguzzi M, Rufer M. A multicomponent family support intervention in intensive care units: study protocol for a multicenter cluster-randomized trial (FICUS Trial). Trials. 2022 Jun 27;23(1):533. doi: 10.1186/s13063-022-06454-y. PMID 35761343
- [Background] Oesch S, Verweij L, Clack L, Finch T, Riguzzi M, Naef R. Implementation of a multicomponent family support intervention in adult intensive care units: study protocol for an embedded mixed-methods multiple case study (FICUS implementation study). BMJ Open. 2023 Aug 8;13(8):e074142. doi: 10.1136/bmjopen-2023-074142. PMID 37553195
- [Derived] Naef R, Jeitziner MM, Riguzzi M, von Felten S, Verweij L, Rufer M, Safford J, Sutter S, Bergmann-Kipfer B, Betschart U, Boltshauser S, Brulisauer N, Brunner C, Buhler PK, Burkhalter H, Dullenkopf A, Heise A, Hertler B, Hoffmann JE, Karde C, Keller Y, Kohler S, Lussmann F, Massarotto P, Moser M, Pietsch U, Segalada DL, Siegrist E, Steiger P, Ruch N, von Dach C, Wenzler MS, Wiegand J, Zante B, Filipovic M; FICUS Study Group. Nurse-Led Family Support Intervention for Families of Critically Ill Patients: The FICUS Cluster Randomized Clinical Trial. JAMA Intern Med. 2025 Sep 1;185(9):1138-1149. doi: 10.1001/jamainternmed.2025.3406. PMID 40720110
- [Derived] von Felten S, Filipovic M, Jeitziner MM, Verweij L, Riguzzi M, Naef R. Multicomponent family support intervention in intensive care units: statistical analysis plan for the cluster-randomized controlled FICUS trial. Trials. 2024 Aug 28;25(1):568. doi: 10.1186/s13063-024-08351-y. PMID 39198900
- See also: Project database of the Swiss National Science Fund (SNSF) — https://data.snf.ch/grants/grant/198778